CLINICAL TRIAL: NCT04676061
Title: Effects of a Progestin on Frequent and/or Prolonged Bleeding With Nexplanon™; a Randomized Double-Blinded Placebo-Controlled Trial
Brief Title: Effects of a Progestin on Frequent and/or Prolonged Bleeding With Nexplanon™
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: It was in the best interest of the investigator to terminate the study earlier than anticipated.
Sponsor: Baylor Research Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 020-291
Record Dates: First submitted 2020-12-11; First posted 2020-12-19 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2023-03

CONDITIONS: Birth Control; Contraception; Implant; Breakthrough Bleeding; Uterine Bleeding
Keywords: Uterine Hemorrhage; Norethindrone Acetate; Contraceptives
MeSH Terms: conditions — Metrorrhagia; Uterine Hemorrhage | interventions — Norethindrone Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control Group (Placebo Comparator): Placebo to Norethindrone acetate (NTA)
  Interventions: Drug: Placebo
- Treatment Group (Active Comparator): Norethindrone acetate (NTA)
  Interventions: Drug: Norethindrone acetate (NTA)

INTERVENTIONS:
Drug: Norethindrone acetate (NTA) — norethindrone acetate, 5 mg tablet, orally, once daily for 7 consecutive days, every 4 weeks
  Arms: Treatment Group
Drug: Placebo — Placebo, tablet, orally, once daily for 7 consecutive days, every 4 weeks
  Arms: Control Group

SUMMARY:
Effects of norethindrone acetate (NTA) in patients with Nexplanon.

DETAILED DESCRIPTION:
The purpose of this study is to find out what effects norethindrone acetate (NTA) has on the duration and recurrence of frequent and/or prolonged bleeding associated with Nexplanon™.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-48
* Between ages of 14-17 with parental/guardian permission
* Women desiring placement of Nexplanon™
* Willing to keep a daily symptom calendar
* Keep appointments
* Women not desiring to become pregnant in the next 2 years

Exclusion Criteria:

* Known or suspected Pregnancy
* Less than 8weeks postpartum
* Menarche less than two years ago
* Current or past history of thrombosis or thromboembolic disorders
* Hepatic tumors (benign or malignant)
* Active liver disease
* Undiagnosed abnormal genital bleeding
* Undiagnosed headaches
* Known or suspected carcinoma of the breast or personal history of breast cancer
* Hypersensitivity to any of the components in Nexplanon™
* BMI greater than 40
* Depomedroxyprogesterone acetate injection in the previous 12 weeks

Ages: 14 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 51 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Number of days of bleeding and spotting | 30 days
  To evaluate days of bleeding and spotting within 90-day intervals by quantifying a self-perception of amount of bleeding on a scale of 0 to 4 and associated symptoms on a scale of 0 to 10 using the Daily Dairy of Symptoms

SECONDARY OUTCOMES:
Quality of life measurements | 30 days
  To evaluate quality of life by comparing the treatment and placebo groups' associated symptoms on a scale of 0 to 10 using the Daily Diary of Symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Stacey, MD, Principal Investigator — Baylor Reserach Institute
Locations (1):
- Baylor Research Institute, Temple, Texas, United States

IPD SHARING:
Plan to Share IPD: No